CLINICAL TRIAL: NCT06414265
Title: Reduction or Elimination of Mitral Regurgitation With the SATURN Trans-Septal TMVR System in Patients With Severe Symptomatic Mitral Regurgitation - CASSINI-EU Trial
Brief Title: Reduction of Mitral Regurgitation With the SATURN Trans-Septal Transcatheter Mitral Valve Replacement (TMVR) System in Patients With Severe Symptomatic Mitral Regurgitation
Acronym: CASSINI-EU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnovHeart (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0181
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): SATURN Trans-septal Transcatheter mitral valve replacement (TMVR) System
  Interventions: Device: Transcatheter mitral valve replacement

INTERVENTIONS:
Device: Transcatheter mitral valve replacement — The SATURN TS TMVR System will be implanted through a transcatheter approach in patients with symptomatic mitral regurgitation.

SUMMARY:
The goal of this clinical trial is to evaluate feasibility, safety, and performance of the SATURN TS TMVR System for the treatment of moderate-to-severe or severe, symptomatic mitral regurgitation through a transcatheter approach. The main questions it aims to answer are:

* is the use of the device feasible?
* is it safe (defined as freedom from device-related major adverse events at 30 days)?
* does it perform (defined as reduction of MR Grade to ≤ 1+ at 30 days)?

Participants will need to do the following as part of the clinical trial:

* complete 6-Minute Walking Test
* complete Quality of Life Questionnaires
* undergo blood evaluations
* CT scan
* 12 lead ECG
* Transesophageal Echocardiography
* Transthoracic Echocardiogram
* the study procedure (valve implantation, right heart catheterization, left arterial pressure, fluoroscopy/ angiogram)

DETAILED DESCRIPTION:
The SATURN Trans-Septal Transcatheter Mitral Valve Replacement System (SATURN TS System) is intended for use in adult patients suffering from heart failure symptoms (NYHA class II or greater) with moderate to severe or severe mitral regurgitation (MR ≥3+) who are deemed to be at high risk for open-heart mitral valve surgery by a multidisciplinary Heart Team including at least a cardiac surgeon and a cardiologist, experienced in the care of patients with mitral valve disease.

CASSINI-EU is a single-arm, prospective, multicenter pilot trial. The purpose of the study is to evaluate feasibility, safety, and performance of the SATURN TS TMVR System for the treatment of moderate-to-severe or severe, symptomatic mitral regurgitation through a transcatheter approach.

Primary objectives are to evaluate the feasibility, safety and performance of the SATURN TS TMVR System at 30 days. Secondary objectives and additional outcomes are long term safety and performance of the SATURN TS TMVR System.

Up to 30 patients will be treated at up to 6 qualified investigational sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older.
2. Symptomatic moderate to severe or severe functional mitral regurgitation (≥ Grade 3+).
3. NYHA functional Class ≥ II. If Class IV, patient must be ambulatory.
4. Ability to tolerate oral anticoagulation.
5. Ability to qualify for bailout surgery (which may include open heart surgery).
6. High risk for open-heart mitral valve surgery due to age, co-morbidities or frailty, as determined by the Heart Team.
7. Willing and able to complete study-related assessments and questionnaires.

Exclusion Criteria:

General Exclusion Criteria

1. Degenerative (i.e. intrinsic valve lesions) mitral regurgitation.
2. Excessive frailty or comorbid conditions that preclude the anticipated benefit of the mitral valve replacement.
3. Life expectancy <1 year due to noncardiac conditions.
4. Endocarditis in the 3 months prior to procedure date.
5. Current admission with acute heart failure exacerbation.
6. Dependency on inotropic agents or mechanical circulatory support.
7. Untreated clinically significant CAD.
8. Active systemic infection.
9. Modified Rankin Scale ≥4 disability.
10. Chronic renal failure defined as eGFR <30 mL/min/m2 or on renal replacement therapy.
11. Severe pulmonary arterial hypertension (PAH), defined as PASP > 60mmHg.
12. Platelets < 90,000.
13. COPD 2 on home oxygen therapy deemed too high risk for intubation.
14. Refuses blood transfusions.
15. Documented bleeding or coagulation disorders (hypo- or hyper-coagulable states).
16. Severe connective tissue disease under chronic immunosuppressive or cortisone therapy.
17. Participating in other investigational studies likely to confound the results or affect the study.
18. Unable or does not sign the study informed consent form.
19. Patients classified as "vulnerable patients" 3 .

    Cardiovascular Exclusion Criteria
20. Myocardial infarction during prior 30 days.
21. Stroke or TIA during prior 90 days.
22. Severe extracardiac arteriopathy (safety measure for extra-circulatory support if surgical conversion is needed).
23. Prior mitral valve treatment (e.g., valve repair or replacement, MitraClip, etc.), and/or anticipated mitral valve treatment prior to enrollment.
24. Prior surgical mechanical valve AVR.
25. Prior TAVI.
26. Need for any planned cardiovascular surgery or intervention (other than for MV disease) within 30 days post-index procedure.
27. CRT or ICD implanted in previous 30 days.
28. Cardiogenic shock, hemodynamic instability, Systolic Blood Pressure <90mmHg, Inotropic dependent or requiring IABP/mechanical circulatory support.
29. CABG or PCI within previous 30 days.
30. Inadequately treated for cardiac condition per applicable standards, such as for coronary artery disease, left ventricular dysfunction, mitral regurgitation, or heart failure, as reviewed by the Patient Screening Committee.
31. Prior or planned heart transplantation (UNOS status 1).
32. Physical evidence of right-sided congestive heart failure:

    1. Patients with ascites.
    2. Patients with anasarca (generalized edema / hydropsy).
33. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or other structural heart disease causing heart failure with the exception of dilated ischemic or non-ischemic cardiomyopathy.

    Procedural Exclusion Criteria
34. Known hypersensitivity or contraindication to procedural or post-procedural medication (e.g., contrast solution, anticoagulation therapy).
35. Documented hypersensitivity to nickel or titanium.
36. Contraindications to TEE imaging

    Cardiac Imaging Exclusion Criteria
37. Left ventricular EF ≤ 30% by echocardiogram.
38. Severe mitral annular calcification, severe mitral stenosis, valvular vegetation or mass.
39. Extensive mitral flail leaflets
40. Evidence of new or untreated intracardiac thrombus, mass, or vegetation.
41. Severe right ventricular dysfunction.
42. Severe tricuspid regurgitation.
43. Hemodynamically significant inter-atrial shunt (ASD).
44. Severe aortic regurgitation or aortic stenosis.
45. Anatomic ineligibility for SATURN TS Bioprosthetic System or SATURN TS procedure as determined by the Screening Committee.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - Freedom from Device Related Major Adverse Events | 30 days post-procedure
  Freedom from device-related major adverse events
Technical Procedural Success Endpoint | Procedure
  Technical success defined as alive patient at exit from procedure room with all the following:
  * Successful access, delivery of the SATURN TS Bioprosthesis, and retrieval of the TS Delivery Systems
  * Correct positioning of the first intended SATURN TS Bioprosthesis
  * Freedom from emergency surgery or mitral valve re-intervention related to the device or access procedure
Efficacy Endpoint - Reduction of Mitral Regurgitation Grade to ≤ 1+ | 30 days post-procedure
  Reduction of MR Grade to ≤ 1+

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Denti, MD, Principal Investigator — San Raffaele Hospital
Locations (3):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No